CLINICAL TRIAL: NCT06592287
Title: Prospective, Dual Arm, Open Ib/II Phase Clinical Study of the Combination of Adebrelimab, Apatinib, and Lrinotecan Liposome for Second-line Treatment of Advanced Gastric Cancer
Brief Title: The Combination of Adebrelimab, Apatinib, and Lrinotecan Liposome for Second-line Treatment of Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xianglin Yuan (Other)
Responsible Party: Sponsor-Investigator, Xianglin Yuan, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-016
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Gastric Cancer
Keywords: Second line advanced gastric cancer; Lrinotecan liposome; Immune checkpoint inhibitors; Anti-L1 antibody; apatinib
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frontline has received treatment with immune checkpoint inhibitors (Experimental): Previously received first-line treatment with immune checkpoint inhibitors, and first-line PFS>7m
  Adebrelimab 1200 mg, iv. q3w
  Apatinib 250 mg po qd
  Lrinotecan liposome 80mg/m2, iv. q3w
  Continue medication until disease progression, toxicity intolerance, initiation of new anti-tumor treatment, withdrawal of knowledge, or continuous medication for at least 2 years.
  Interventions: Drug: Adebrelimab + Apatinib + Lrinotecan liposome
- Previously not received immune checkpoint inhibitor treatment (Experimental): those who have received standard systemic chemotherapy
  Adebrelimab 1200 mg, iv. q3w
  Apatinib 250 mg po qd
  Lrinotecan liposome 80mg/m2, iv. q3w
  Continue medication until disease progression, toxicity intolerance, initiation of new anti-tumor treatment, withdrawal of knowledge, or continuous medication for at least 2 years.
  Interventions: Drug: Adebrelimab + Apatinib + Lrinotecan liposome

INTERVENTIONS:
Drug: Adebrelimab + Apatinib + Lrinotecan liposome — Adebrelimab 1200 mg, iv. q3w
  Apatinib 250 mg po qd
  Lrinotecan liposome 80mg/m2, iv. q3w
  Continue medication until disease progression, toxicity intolerance, initiation of new anti-tumor treatment, withdrawal of knowledge, or continuous medication for at least 2 years.

SUMMARY:
This study is a prospective, dual arm, open Ib/II phase clinical trial, with the main objective of exploring the safety and efficacy of Adebrelimab combined with Apatinib and Lrinotecan liposome for second-line treatment of advanced gastric cancer.

The study is divided into two stages. The first stage is the safety introduction period, which includes 6 patients. Observe whether the subjects experience dose limiting toxicity (DLT) during the observation period. If no subjects experience DLT during the observation period, the study enters the next stage. The dose of Lrinotecan liposome used during the safety introduction period is 80mg/m2, and the DLTs observation period is 1 cycle. If the patient cannot tolerate it, the dose will be reduced to 60mg/m2.

In the second stage, advanced gastric cancer subjects who have progressed to first-line treatment will be included in two cohorts: those who have previously received immune checkpoint inhibitor therapy and have first-line PFS>7m (cohort 1) and those who have received standard systemic chemotherapy (cohort 2). 30 subjects will be included in each population, and a total of 66 subjects are planned to be enrolled.

The study includes a screening period (from the signing of the informed consent form by the subjects to the first treatment, not exceeding 28 days), a treatment period (Adebrelimab combined with Apatinib and Lrinotecan liposome), and a follow-up period (including safety and survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 to 75 years old, both male and female are acceptable;
2. Patients with gastric adenocarcinoma or gastroesophageal junction adenocarcinoma diagnosed by histology or cytology;
3. Patients who have only received one failed systemic treatment for advanced diseases in the past; After undergoing immunotherapy, the PFS of the treatment regimen containing immune checkpoint inhibitors must be greater than 7 months;
4. According to the evaluation criteria for solid tumor efficacy 1.1 (RECIST v1.1), there should be at least one measurable lesion that has not received local treatment such as radiotherapy (lesions located within the previously irradiated area can also be selected as target lesions if progression is confirmed);
5. ECOG score: 0-1 point;
6. Expected survival period ≥ 12 weeks;
7. The main organ functions well and the laboratory test data meets the following standards: (1) Blood routine: absolute neutrophil count ≥ 1.5 × 109/L (or greater than the lower limit of normal laboratory values in the research center), platelet count ≥ 100 × 109/L, hemoglobin ≥ 90g/L; (2) Liver function: serum total bilirubin ≤ 1.5 times the upper limit of the standard value (ULN), AST and ALT ≤ 2.5 times ULN. If the patient has liver metastasis, this standard is ≤ 5 times ULN; (3) Renal function: CrCl ≥ 60 ml/min/1.73 m2 (calculated according to the Cockcroft Gault formula);
8. Female subjects with fertility, as well as male subjects with partners who are fertility women, are required to use a medically approved contraceptive measure (such as intrauterine devices, birth control pills, or condoms) during the study treatment period, at least 6 months after the last use of Adebrelimab, at least 6 months after the last use of Apatinib, and at least 6 months after the last use of chemotherapy;
9. HER2 negative;
10. Voluntarily join this study, sign informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. History of gastrointestinal perforation and/or fistula within 6 months prior to the first use of medication;
2. There is uncontrollable pleural effusion, pericardial effusion, or peritoneal effusion that requires repeated drainage;
3. Have a history of allergies to any component of Adebrelimab in the past;
4. Have received any of the following treatments:

   1. Received any other investigational drug within 4 weeks prior to the first use of the investigational drug or had a half-life of no more than 5 from the last investigational drug;
   2. Simultaneously enrolled in another clinical study, unless it is an observational (non interventional) clinical study or an interventional clinical study follow-up;
   3. Received anti-tumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, or tumor embolization) within 2 weeks prior to the first use of the investigational drug;
   4. Subjects who need to receive corticosteroids (equivalent to>10mg prednisone per day) within 2 weeks prior to the first use of the study drug. Allow the use of hormones for routine chemotherapy pretreatment without the need for dose adjustment. Other special circumstances require communication with the researcher. In the absence of active autoimmune diseases, inhalation or local use of steroids and corticosteroids with a dosage greater than 10mg/day of prednisone efficacy dose are allowed as substitutes for adrenal cortex hormones;
   5. Individuals who have received anti-tumor vaccines or have received live vaccines within 4 weeks prior to the first administration of the study drug;
   6. Having undergone major surgery or suffered severe trauma within 4 weeks prior to the first use of the investigational drug;
5. The toxicity of previous anti-tumor treatments has not recovered to ≤ CTCAE 5.0 Grade 1 (excluding hair loss) or the level specified in the inclusion/exclusion criteria;
6. Patients with active central nervous system metastases;
7. Active autoimmune diseases, history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to the above diseases or syndromes); Excluding childhood asthma/allergies with vitiligo or those who have already recovered, patients who do not require any intervention in adulthood; Autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with a stable dose of insulin;
8. Have a history of immune deficiency, including HIV test positive, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation, or active hepatitis (hepatitis B reference: HBV DNA test value exceeds 500 IU/ml or 2500 copies/mL);
9. The subject has uncontrolled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year; (4) Clinically significant supraventricular or ventricular arrhythmias that have not been clinically intervened or are still poorly controlled after clinical intervention;
10. Within 4 weeks prior to the first use of the investigational drug, there has been a severe infection (CTCAE 5.0>grade 2), such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc; Baseline chest imaging examination suggests the presence of active pulmonary inflammation, symptoms and signs of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, except for prophylactic use of antibiotics;
11. History of interstitial lung disease (excluding history of radiation pneumonia and non infectious pneumonia that have not been treated with steroids);
12. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within the past year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than one year ago but without formal treatment;
13. Diagnosed with any other malignant tumor within 5 years prior to the first use of the investigational drug, except for malignant tumors with low-risk metastasis and mortality risk (5-year survival rate>90%), such as basal cell or squamous cell carcinoma or cervical carcinoma in situ that have been adequately treated;
14. Pregnant or lactating women;
15. According to the researcher's assessment, there may be other factors that could force the subject to terminate the study midway, such as having other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival（PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months

SECONDARY OUTCOMES:
Median overall survival (mOS) | From date of randomization until date of death from any cause, assessed up to 12 months
Objective response rate (ORR) | From enrollment to initial efficacy evaluation，Expected to be evaluated in about 2 months
Disease Control Rate（DCR） | From enrollment to initial efficacy evaluation，Expected to be evaluated in about 2 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From enrollment to 90 days after the last medication

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided